CLINICAL TRIAL: NCT03045757
Title: Evaluating Oral Motor Skills of Neonates Requiring Congenital Heart Surgery and the Impact on Oral Feeding Readiness
Brief Title: Evaluating Dysphagia in Neonates With CHD
Status: Terminated | Type: Observational
Why Stopped: Dr. Fogel left the organization, and no other clinician was available to continue the study. Data was never collected for the study.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 6540; K5900376 (Other: Advocate Health Care)
Record Dates: First submitted 2017-01-26; First posted 2017-02-07 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia of Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Newborn: Healthy Newborn
- CHD Neonates: Neonates born with CHD before and after surgical repair

SUMMARY:
The overall goal of this study is to describe the oral motor skills of neonates born with congenital heart defects, both before and after cardiac surgery, and to evaluate current measures of feeding motor skills and feeding readiness in this population using the Neonatal Oral Motor Assessment Scale (NOMAS) and the Infant Driven Feeding Scale.

The specific aims are to:

1. Describe the oral motor skills of infants with CHD before surgery as compared with normal full-term newborn (>37 weeks) using the NOMAS
2. Describe the oral motor skills of infants with CHD after surgery as compared with those same infants before surgery using the NOMAS.
3. Determine if the current Infant Driven Feeding Readiness Scale appropriately identifies which children with CHD are ready for oral feeding. (A. Feeding Readiness Scale, B. Quality of Nippling Scale at the 1st post- operative feeding evaluation)
4. Describe the unique characteristics of oral motor skills in infants with CHD (ie. Wide jaw excursions, poor latch, etc.) Our hypothesis is that infants with CHD will have dysfunctional sucking patterns before surgical repair as compared to normal newborns. This dysfunctional sucking pattern in infants with CHD will have worsened post-surgery as compared to pre-surgery. In addition, the Infant Driven Feeding Scale will be utilized to predict that many infants with CHD will not be ready for oral feedings, however most of those patients will go on to successfully take oral feedings.

ELIGIBILITY:
Inclusion Criteria:

* Full-term newborns with normal physical exam that are delivered > 37 weeks gestation (healthy newborn arm).

or

* Newborn with CHD born > 37 weeks gestation, are hemodynamically stable and who require surgical correction in the first 30 days of life (CHD arm).

Exclusion Criteria:

* Full-term newborn arm
* Newborn admitted into the NICU
* Genetic syndromes
* Congenital abnormalities or signs of developmental delay

  · Infants with CHD arm
* Newborn requiring intubation prior to evaluation (Note: Infants with CHD with genetic or other malformations not specifically mentioned will not be excluded due to their prevalence in this population)
* Down Syndrome
* Trisomy 13, Trisomy 18
* Congenital anomalies of facial structure or musculature specifically cleft lip, hard or soft palate

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy newborns and neonates with CHD
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Oral motor skills of infants with CHD utilizing the NOMAS | 1 year
Type and quality of oral motor skills of infants with CHD before cardiothoracic surgery as measured by NOMAS | 1 year
Type and quality of feeding readiness using the Infant Driven Feeding Scales with infants with CHD after cardiothoracic surgery | 1 year
Type and Quality of oral motor skills in newborn infants as measured by NOMAS | 1 year
Type and quality of oral motor skills of infants with CHD after cardiothoracic surgery as measured by NOMAS | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Fogel, MSCCC-SLP/L, Principal Investigator — Advocate Healthcare
Locations (1):
- Advocate Children's Hospital, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No